CLINICAL TRIAL: NCT00000926
Title: Phase III Nonoxynol-9 and HIV Infection
Brief Title: A Study of Nonoxynol-9 (N-9) and HIV Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: Double | Purpose: Prevention
Other Study IDs: HIVNET 016 Pilot; 11712 (Registry Identifier: DAIDS ES); HIVNET 016
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Nonoxynol
MeSH Terms: conditions — HIV Infections | interventions — Nonoxynol

INTERVENTIONS:
Drug: Nonoxynol-9

SUMMARY:
The purpose of this study is to see if nonoxynol-9 (N-9) gel used in the vagina can prevent the spread of HIV.

Most of the people with HIV in the world today live in southern Africa. Because this population is not likely to use condoms, an HIV-prevention method that women can control is needed. N-9 used in the vagina may help prevent the spread of HIV and other sexually transmitted diseases.

DETAILED DESCRIPTION:
Intravaginal application of N-9 may help protect women from HIV and other STD infection. Low rates of condom use in sub-Saharan African populations, which constitute the majority of HIV infections, dictate the need for prophylactic methods women can control.

This trial will be conducted in Zimbabwe and Malawi. The Phase III trial is preceded by a 2-week safety and acceptability pilot study to determine the extent of genital irritation caused by N-9 and the placebo. Following the pilot study and prior to screening for enrollment in the Phase III trial, potential volunteers will participate in a 2-month behavioral counseling program that will encourage the use of condoms. Only participants who decide they cannot or will not be consistent condom users are enrolled in the main study. Study participants are given N-9 gel or placebo to use each time they have vaginal sexual intercourse for 18 to 36 months. Participants have a follow-up evaluation once a month; a pelvic exam and blood tests are performed every third month.

ELIGIBILITY:
Inclusion Criteria

Volunteers may be eligible if they:

* Are HIV-negative.
* Are sexually active and expect to have vaginal intercourse at least twice a week during the study.
* Are willing to keep a diary of their sexual behavior and N-9 use.
* Are willing to have regular clinic visits including pelvic exams.
* Are at least 18 years old.
* Are female.

Exclusion Criteria

Volunteers will not be eligible if they:

* Have had a child or an abortion in the past 42 days.
* Are allergic to latex or N-9.
* Have genital sores.
* Have syphilis, chlamydia, gonorrhea, or trichomoniasis.
* Are enrolled in another study for a product like N-9.
* Expect to use another vaginal product other than N-9 during the study.
* Are pregnant.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4400
Dates: Study Completion 2001-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Taha E.Taha, Study Chair; Nancy Padian, Study Chair
Locations (1):
- Julia Welch, Research Triangle Park, North Carolina, United States

REFERENCES:
- [Result] Kumwenda N, Hoffman I, Chirenje M, Kelly C, Coletti A, Ristow A, Martinson F, Brown J, Chilongozi D, Richardson B, Rosenberg Z, Padian N, Taha T. HIV incidence among women of reproductive age in Malawi and Zimbabwe. Sex Transm Dis. 2006 Nov;33(11):646-51. doi: 10.1097/01.olq.0000223283.27142.9f. PMID 16773032